CLINICAL TRIAL: NCT00382265
Title: Study of Tamsulosin for Urolithiasis in the Emergency Department
Brief Title: Tamsulosin for Urolithiasis in the Emergency Dept
Acronym: STONE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrew Meltzer (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Andrew Meltzer, Principal Investigator, George Washington University
Organization: George Washington University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RO1 DK71603; U01DK096037 (NIH); U01DK071603 (NIH); U34DK090957 (NIH)
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-11

CONDITIONS: Ureterolithiases
Keywords: urolithiasis; renal colic; kidney stones; urinary stone disease
MeSH Terms: conditions — Ureterolithiasis; Urolithiasis; Renal Colic; Kidney Calculi | interventions — Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tamsulosin (Active Comparator): Tamsulosin 0.4mg PO qd for 28 days
  Interventions: Drug: tamsulosin
- Placebo (Placebo Comparator): Placebo PO qd for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: tamsulosin — tamsulosin 0.4mg po qd for 28 days
  Arms: Tamsulosin
Other: Placebo — placebo po qd for 28 days
  Arms: Placebo

SUMMARY:
Urolithiasis is a disease that effects 12% of the population and its incidence is growing. In the US there are over 1.1 million visits annually to Emergency Departments for renal colic. The disease is extremely painful, often requiring large amounts of narcotic analgesia, and results in lost work days. Moreover, up to 30% of patients may eventually require lithotripsy or surgical removal of the stone. Currently there are no medical interventions other than analgesia which are offered to patients.

Based on encouraging results from several small European clinical studies, the researchers hypothesize that the administration of tamsulosin to patients with symptomatic urolithiasis will enhance stone passage, and reduce both the time to recovery and the need for surgical intervention or lithotripsy. The researchers will conduct a study by identifying and recruiting patients presenting with urolithiasis in the emergency departments of four institutions.

A total of 500 consenting subjects will be randomly assigned to one of two groups:

1. tamsulosin for a maximum of 28 days;
2. placebo for a maximum of 28 days.

In addition, both groups will receive standard analgesic therapy.

The study team, which will be blinded to treatment status, will monitor each subject's clinical progress and outcome. The primary objectives of this study are:

1. to determine if tamsulosin is effective, and
2. to evaluate the safety of the therapy.

Another objective is to identify the most appropriate clinical subgroup(s) for treatment.

If the therapeutic benefits observed in smaller clinical studies are replicated, administration of these medications should produce several benefits, including:

1. a reduction in time to pain free recovery and hence a more rapid return to employment;
2. decreased requirements for narcotic analgesia;
3. less need for urological out-patient clinic follow-up;
4. decreased need for surgical intervention or lithotripsy; and
5. substantial cost savings.

If this therapy is beneficial, it will represent a major advance in the treatment of urolithiasis. This objective is a major stated goal of the NIDDK (National Institute of Diabetes and Digestive and Kidney Diseases) Clinical Urology Program, which has a stated mission to improve the treatment of urolithiasis.

Kidney stones are a major public health issue, and one person in eight will be affected by the disease. If the hypothesis is verified, the researchers will provide the first medical therapy ever for this disease. This therapy, if effective, will reduce the amount of time a patient is off work because of the pain from the disease, and may also reduce the need for expensive and time-consuming surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Evidence of ureterolithiasis (i.e. stone is located in ureter, not in bladder) as demonstrated on radiographic studies, specifically non-contrast spiral CT.
3. Willingness to participate and able to proceed with standard outpatient management (no personal or job-related issues, e.g. airline pilot.
4. Has a telephone in order to be contacted for follow-up.

Exclusion Criteria:

1. Patient desiring or requiring immediate surgical intervention making then not a candidate for outpatient kidney stone management.
2. Current urinary tract infection based on urine dipstick as admission and urgent procedural management are likely indicated.
3. Known anatomical genitourinary abnormalities or prior Genitourinary surgeries.
4. Positive pregnancy test making proper radiological imaging contraindicated.
5. Breastfeeding mothers.
6. History of hypersensitivity to tamsulosin.
7. Current use of alpha blockers or calcium channel blockers.
8. Current use of steroids which may have an independent effect on stone expulsion.
9. Spontaneous stone expulsion prior to enrollment.
10. Largest stone dimension ≥ 9mm assessed using radiologic imaging, being very unlikely to pass spontaneously.
11. Presence of stone in the bladder.
12. Current use of vardenafil which is tamsulosin contraindicated.
13. Ipsilateral, transplanted or solitary kidney as hospitalization may be necessary.
14. Known renal insufficiency.
15. Fever defined as >101.5°F which may indicate infection.
16. Floppy iris syndrome which is tamsulosin contraindicated.
17. Planned cataract surgery in the next 60 days which is tamsulosin contraindicated.
18. Prisoners /wards of state.
19. Prior enrollment in STONE (Candidates who are screened and found ineligible may be rescreened at a later date.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2008-01; Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Meltzer, MD, Principal Investigator — The George Washington University
Locations (4):
- United States (4):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Meltzer AC, Wolfson AB, Mufarrij P, MacPherson C, Montano N, Kirkali Z, Burrows PK, Jackman SV. Analgesic and Opioid Use for Patients Discharged from the Emergency Department with Ureteral Stones. J Endourol. 2021 Jul;35(7):1067-1071. doi: 10.1089/end.2020.0835. Epub 2021 Jan 21. PMID 33213185
- [Derived] Meltzer AC, Burrows PK, Wolfson AB, Hollander JE, Kurz M, Kirkali Z, Kusek JW, Mufarrij P, Jackman SV, Brown J. Effect of Tamsulosin on Passage of Symptomatic Ureteral Stones: A Randomized Clinical Trial. JAMA Intern Med. 2018 Aug 1;178(8):1051-1057. doi: 10.1001/jamainternmed.2018.2259. PMID 29913020
- [Derived] Burrows PK, Hollander JE, Wolfson AB, Kurz MC, Richards L, DiFiore S, Watts P, Patkar N, Brown J, Jackman S, Kirkali Z, Kusek JW, Michel C, Meltzer AC; STONE Study Investigators. Design and challenges of a randomized clinical trial of medical expulsive therapy (tamsulosin) for urolithiasis in the emergency department. Contemp Clin Trials. 2017 Jan;52:91-94. doi: 10.1016/j.cct.2016.11.010. Epub 2016 Nov 23. PMID 27890522

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator:1: Tamsulosin 0.4mg PO
  tamsulosin: tamsulosin 0.4mg po qd for 28 days
- Placebo Comparator:2: Placebo
  tamsulosin: tamsulosin 0.4mg po qd for 28 days
Period: Overall Study
Arm/Group | Active Comparator:1 | Placebo Comparator:2
Started | 267 | 245
Completed | 258 | 239
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Tamsulosin Group: Tamsulosin 0.4mg PO
  tamsulosin: tamsulosin 0.4mg po qd for 28 days
- Placebo Group: Placebo for 28 days
- Total: Total of all reporting groups
Arm/Group | Tamsulosin Group | Placebo Group | Total
Number analyzed (Participants) | 267 | 245 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.6) | 39.3 (12.9) | 40.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 139
  Male | 197 | 176 | 373
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-White Race | 56 | 54 | 110
Region of Enrollment [Number; unit: participants]
  United States | 267 | 245 | 512

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Passing Their Stone Within 28 Days by Self Report
Description: Hypothesis: The administration of tamsulosin after the clinical and radiographic diagnosis of acute urolithiasis will produce an increase in the proportion of patients passing their stone within 28 days.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Tamsulosin: Tamsulosin 0.4mg PO
  tamsulosin: tamsulosin 0.4mg po qd for 28 days
- Placebo: Placebo
  tamsulosin: tamsulosin 0.4mg po qd for 28 days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 258 | 239
Participants | 128 | 113

2. Secondary Outcome: Any Pain Medication
Description: Patients on any pain medication at day 28
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo pill po qd for 28 days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 226 | 210
Participants | 22 | 24

3. Secondary Outcome: Need for Surgical Intervention
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo Pill qd for 28 days
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 214 | 189
Participants | 14 | 13

4. Secondary Outcome: Crossover to Open Label Tamsulosin
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 214 | 189
Participants | 15 | 14

5. Secondary Outcome: Confirmation of Stone Passage on CT
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Tamsulosin | Placebo
Number analyzed (Participants) | 122 | 116
Participants | 102 | 90

6. Secondary Outcome: Return to Work (if Employed)
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Placebo pill po qd for 28 days
Arm/Group | Tamsulosin | Control Group
Number analyzed (Participants) | 204 | 188
Participants | 202 | 185

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 90 days after each patient enrollment in the study.
Arm/Group | Tamsulosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/267 | 0/245
Serious Adverse Events (participants affected / at risk) | 0/267 | 0/245
Other Adverse Events (participants affected / at risk) | 0/267 | 0/245

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT00382265/Prot_SAP_ICF_000.pdf